CLINICAL TRIAL: NCT05923008
Title: A Phase 1/2, Multicenter, Open-label Study of IBI130 in Subjects With Unresectable, Locally Advanced or Metastatic Solid Tumors
Brief Title: A Clinical Study of IBI130 for Subjects With Unresectable, Locally Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI130A101
Record Dates: First submitted 2023-06-19; First posted 2023-06-28 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBI130 (Experimental): IBI130
  Interventions: Drug: IBI130

INTERVENTIONS:
Drug: IBI130 — Subjects will receive IBI130 until unacceptable toxicity, disease progression, withdrawal of consent, occurrence of other reasons for discontinuing study therapy, or for a maximum of 24 months of treatment, whichever occurs first.

SUMMARY:
This is a phase 1/2 multicenter, open-label, first-in-human study of IBI130. It includes a phase 1 dose escalation and expansion section to identify MTD/RP2D of IBI130, plan to enroll 20~182 subjects,and a phase 2 to explore efficacy, safety and tolerability of IBI130 at RP2D in specified types of solid tumor.Approximately 150 evaluable subjects will be enrolled for phase 2.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with the ability to understand and give written informed consent for participation in this trial, including all evaluations and procedures as specified by this protocol;
2. Male or female subjects ≥ 18 years old;
3. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1;
4. Anticipated life expectancy of ≥ 12 weeks;
5. Adequate bone marrow and organ function

Exclusion Criteria:

1. Enrolled in any other interventional clinical research except unless only involved in an observational study (non-interventional) or in the follow-up phase of an interventional study;
2. Received previous anti-tumor therapy within 4 weeks or 5 half-lives of the anti-tumor regimens before the first administration of study drug, whichever is shorter;
3. Plan to receive other antitumor therapy during the study excluding palliative radiotherapy for the purpose of symptom (like pain) relief that must also do not have impact on tumor assessment throughout the study;
4. Received live vaccines within 4 weeks prior to first administration of the study drug or plan on receiving any live vaccine during the study;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2023-11-14 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) | Up to 30 days post last dose
  Adverse events will be assessed by investigator(s) according to NCI-CTCAE v5.0

SECONDARY OUTCOMES:
objective response rate (ORR) | Time from first dose to best response to treatment, assessed up to 3 years
  ORR is the percentage of complete response(CR) plus partial response assessed(PR) per RECIST v1.1 criteria
duration of response(DoR) | Duration of response from the first documentation of objective response (confirmed CR or PR) to the first documented disease progression, assessed up to 3 years
  For subjects with CR or PR,duration of response(DoR) is the time from the first documented CR or PR to disease progression assessed per RESICT v1.1 criteria or death
overall survival (OS) | Time from first dose to death, assessed up to 3 years
  Time from the date of the first dose to death of the subject due to any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Sunshine Coast University, Birtinya, Queensland, Australia